CLINICAL TRIAL: NCT00516139
Title: Lamotrigine Extended-Release in Elderly Patients With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEP105972
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Epilepsy
Keywords: Epilepsy elderly seizure
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lamotrigine (Experimental): Open-label lamotrigine
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Open-label

SUMMARY:
This study is being conducted to determine the safety and tolerability of lamotrigine (LTG) in elderly patients with epilepsy. This study will be carried out using an extended-release formulation of lamotrigine (LTG-XR) that will allow once-a-day dosing.

ELIGIBILITY:
Inclusion criteria:

* Confident diagnosis of epilepsy
* Currently treated with one or two antiepileptic medications
* Able to complete a seizure diary

Exclusion criteria:

* History of hypersensitivity to lamotrigine
* Progressive diseases that would interfere with the study objectives

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (57):
- United States (57):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullteron, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ponte Vedra Beach, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Suwanee, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Scarborough, Maine
  - GSK Investigational Site, Burlington, Massachusetts
  - GSK Investigational Site, Hopedale, Massachusetts
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Cedarhurst, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Schenectady, New York
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Columbia, Tennessee
  - GSK Investigational Site, Cordova, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Bremerton, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: LEP105972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LEP105972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LEP105972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LEP105972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LEP105972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LEP105972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LEP105972 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 4 phases (Ph): 7-week (w) Dose-escalation Ph, 8-w Adjunctive Maintenance (AM) Ph, 13-w Adj. Optimization (AO) Ph or 13-w Conversion/Monotherapy (C/M) Ph, and a 2-5 w Taper/Follow up (T/F) Ph.
Groups:
- Lamotrigine (LTG)-Extended Release (XR) Tablets: LTG-XR tablets (25, 50, 100, and 200 milligrams [mg]) administered once a day (OD) in the 7-week (w) Dose-Escalation Phase and titrated to target doses of 300, 500, or 200 mg/day for participants (par.) depending on their concomitant antiepileptic drug (AED), followed by an 8-w Adjunctive Maintenance Phase in which LTG-XR tablets were administered OD at the target dose. Par. on a single concomitant AED who converted to LTG-XR monotherapy (based on investigator's judgment) entered the 5-w Conversion Phase, followed by an 8-w Monotherapy Phase, whereas par. who did not transition to monotherapy entered the 13-w Adjunctive Optimization Phase. At the end of the study, par. entered the 2- to 5-w Taper/Follow-Up Phase, in which par. either switched to commercial LTG (received same total daily dose of commercial LTG in 2 divided doses [BID]) or did not switch to commercial LTG (current dose was reduced by approximately one-fourth per week) with a final visit 2 weeks after last LTG-XR dose.
Period: Overall Study
Arm/Group | Lamotrigine (LTG)-Extended Release (XR) Tablets
Started | 122
Completed | 84 (Study completers completed Escalation, AM, and either AO or both Conversion and Monotherapy Phases.)
Not Completed | 38
Not completed — Adverse Event | 27
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 8
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Groups:
- LTG-XR Tablets: LTG-XR tablets (25, 50, 100, and 200 milligrams [mg]) administered once a day (OD) in the 7-week (w) Dose-Escalation Phase and titrated to target doses of 300, 500, or 200 mg/day for participants (par.) depending on their concomitant antiepileptic drug (AED), followed by an 8-w Adjunctive Maintenance Phase in which LTG-XR tablets were administered OD at the target dose. Par. on a single concomitant AED who converted to LTG-XR monotherapy (based on investigator's judgment) entered the 5-w Conversion Phase, followed by an 8-w Monotherapy Phase, whereas par. who did not transition to monotherapy entered the 13-w Adjunctive Optimization Phase. At the end of the study, par. entered the 2- to 5-w Taper/Follow-Up Phase, in which par. either switched to commercial LTG (received same total daily dose of commercial LTG in 2 divided doses [BID]) or did not switch to commercial LTG (current dose was reduced by approximately one-fourth per week) with a final visit 2 weeks after last LTG-XR dose.
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected for the Safety Population, which included all participants who were enrolled and took at least one dose of the study drug. One participant enrolled in the study did not take at least one dose of the study drug.
  Years | 72.5 (5.53)
Gender [Count of Participants; unit: Participants] — Baseline characteristics were collected for the Safety Population, which included all participants who were enrolled and took at least one dose of the study drug. One participant enrolled in the study did not take at least one dose of the study drug.
  Participants
    Female | 59
    Male | 62
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected for the Safety Population, which included all participants who were enrolled and took at least one dose of the study drug. One participant enrolled in the study did not take at least one dose of the study drug. Participants are allowed to select more than one race.
  participants
    African American/African Heritage | 14
    Asian - South East Asian Heritage | 2
    White - Arabic/North African Heritage | 1
    White - White/Caucasian/European Heritage | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Serious Adverse Event (SAE) and Any Non-serious Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or causes its prolongation, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event. A complete list of all SAEs and AEs experienced in the study can be found in the SAE/AE section.
Time Frame: From Baseline (Week 0) until 3 weeks after the end of treatment (Week 30 or 33)
Population: Safety Population: all participants who were enrolled and took at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 121
participants
  Participants with any SAE | 22
  Participants with any non-serious AE | 112

2. Secondary Outcome: Percent Change From Baseline (BL) in Weekly Seizure (sz.) Frequency for All Partial Seizures During Each Phase of the Study
Description: Partial-onset sz. have a focal site of onset; sz. activity is initially limited to 1 brain hemisphere. Partial sz. can remain simple or complex, or evolve to generalized tonic-clonic sz. Participants (par.) recorded the number of sz., by type as well as the episode duration of innumerable sz. activity), in daily diaries. If par. withdrew from study, data were averaged for the study portion the par. completed up to the time of drug discontinuation. Percent change from BL = (BL value minus study phase value divided by BL value) x 100; positive values indicate reduction from BL in sz. frequency.
Time Frame: Baseline (Week 0), Dose-Escalation Phase (Week 7), Maintenance Phase (Week 15), Adjunctive Optimization Phase (Week 28), Conversion Phase (Week 20), Monotherapy Phase (Week 28), and end of treatment (Week 30 or 33)
Population: Safety Population. Only those participants who had seizures at baseline were analyzed.
Measure: Median (Full Range); unit: Percent change in seizure frequency
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 55
Percent change in seizure frequency
  Dose-Escalation Phase (Week 7), n=55 | 97.8 [-146.3 to 100.0]
  Maintenance Phase (Week 15), n=43 | 100.0 [-162.5 to 100.0]
  Adjunctive Optimization Phase (Week 28), n=15 | 100.0 [33.3 to 100.0]
  Conversion Phase (Week 20), n=24 | 100.0 [-44.5 to 100.0]
  Monotherapy Phase (Week 28), n=24 | 100.0 [-269.8 to 100.0]
  End Of Treatment (Week 30/33), n=55 | 90.4 [-86.7 to 100.0]

3. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in Weekly Seizure Frequency During Each Phase of the Study
Description: Participants recorded the number of seizures, by seizure type, as well as the duration of episodes of innumerable seizure activity in their daily diaries during all phases of the study. For participants who withdrew from the study, seizure data were averaged for the portion of the study the participant completed up to the time of study drug discontinuation. Participants who experienced a change from Baseline in the weekly seizure frequency were categorized as having a >=25%, >=50%, >=75%, or 100% reduction or a >=50% increase in percent change from Baseline in weekly seizure frequency.
Time Frame: Baseline (Week 0), Dose-Escalation Phase (Week 7), Maintenance Phase (Week 15), Adjunctive Optimization (Adj O) Phase (Week 28), Conversion Phase (Week 20), Monotherapy Phase (Week 28), and end of treatment (ET, Week 30 or 33)
Population: Safety Population. Only those participants who had seizures at baseline were analyzed.
Measure: Number; unit: participants
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 55
participants
  Dose-Escalation (Week 7), >=25% reduction, n=55 | 49
  Dose-Escalation (Week 7), >=50% reduction, n=55 | 41
  Dose-Escalation (Week 7), >=75% reduction, n=55 | 30
  Dose-Escalation (Week 7), 100% reduction, n=55 | 27
  Dose-Escalation (Week 7), >=50% increase, n=55 | 2
  Maintenance (Week 15), >=25% reduction, n=43 | 39
  Maintenance (Week 15), >=50% reduction, n=43 | 37
  Maintenance (Week 15), >=75% reduction, n=43 | 33
  Maintenance (Week 15), 100% reduction, n=43 | 30
  Maintenance (Week 15), >=50% increase, n=43 | 2
  Adj O (Week 28), >=25% reduction, n=15 | 15
  Adj O (Week 28), >=50% reduction, n=15 | 14
  Adj O (Week 28), >=75% reduction, n=15 | 12
  Adj O (Week 28), 100% reduction, n=15 | 11
  Adj O (Week 28), >=50% increase, n=15 | 0
  Conversion (Week 20), >=25% reduction, n=24 | 23
  Conversion (Week 20), >=50% reduction, n=24 | 23
  Conversion (Week 20), >=75% reduction, n=24 | 19
  Conversion (Week 20), 100% reduction, n=24 | 17
  Conversion (Week 20), >=50% increase, n=24 | 0
  Monotherapy (Week 28), >=25% reduction, n=24 | 23
  Monotherapy (Week 28), >=50% reduction, n=24 | 20
  Monotherapy (Week 28), >=75% reduction, n=24 | 17
  Monotherapy (Week 28), 100% reduction, n=24 | 13
  Monotherapy (Week 28), >=50% increase, n=24 | 1
  ET (Week 30/33), >=25% reduction, n=55 | 47
  ET (Week 30/33), >=50% reduction, n=55 | 44
  ET (Week 30/33), >=75% reduction, n=55 | 36
  ET (Week 30/33), 100% reduction, n=55 | 24
  ET (Week 30/33), >=50% increase, n=55 | 1

4. Secondary Outcome: Number of Seizure-free Participants at Baseline Who Remained Seizure-free Throughout the Entire Treatment Period
Description: Participants were considered to be seizure-free if they did not report any seizures at Baseline.
Time Frame: Week 30 or 33
Population: Safety Population. Participants who were seizure-free at Baseline were analyzed.
Measure: Number; unit: participants
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 66
participants
  Remained Seizure-Free | 53
  Did Not Remain Seizure-Free | 13

5. Secondary Outcome: Number of Participants With Changes From Baseline in Seizure Severity in the Indicated Categories, as Measured by the Investigator's Global Evaluation (IGE) Scale
Description: Investigators rated the participants' seizure severity at Weeks 15 and 28 of the study treatment by using the IGE scale, comprised of 7 categories: 3 for improvement (mild improvement, moderate improvement, and marked improvement), 3 for deterioration (marked deterioration, moderate deterioration, mild deterioration), and 1 for no change. Investigators assessed the degree of the participants' improvement or deterioration or determined whether the participants' condition had not changed compared to their Baseline condition.
Time Frame: Week 15 (Adjunctive Maintenance [Adj M] Phase), Week 28 (Adjunctive Optimization [Adj O] Phase), Week 28 (Monotherapy [Mono] Phase), and Week 28 (Early Withdrawal [WD])
Population: Safety Population. Only those participants who had seizures at baseline were analyzed.
Measure: Number; unit: participants
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 91
participants
  Week 15, Adj M Phase, Improvement, n=91 | 36
  Week 15, Adj M Phase, No change, n=91 | 54
  Week 15, Adj M Phase, Deterioration, n=91 | 1
  Week 28, Adj O Phase, Improvement, n=21 | 13
  Week 28, Adj O Phase, No change, n=21 | 7
  Week 28, Adj O Phase, Deterioration, n=21 | 1
  Week 28, Mono Phase, Improvement, n=63 | 29
  Week 28, Mono Phase, No change, n=63 | 33
  Week 28, Mono Phase, Deterioration, n=63 | 1
  Week 28, WD, Improvement, n=35 | 7
  Week 28, WD, No change, n=35 | 25
  Week 28, WD, Deterioration, n=35 | 3

6. Secondary Outcome: Number of Participants With Changes From Baseline in Overall Clinical Status in the Indicated Categories, as Measured by the IGE Scale
Description: Investigators rated the participants' overall clinical status at Weeks 15 and 28 of the study treatment by using the IGE scale, comprised of 7 categories: 3 for improvement (mild improvement, moderate improvement, and marked improvement), 3 for deterioration (marked deterioration, moderate deterioration, mild deterioration), and 1 for no change. Investigators assessed the degree of the participants' improvement or deterioration or determined whether the participants' condition had not changed compared to their Baseline condition.
Time Frame: as for outcome 5
Population: Safety Population. Participants with missing data were not analyzed.
Measure: Number; unit: participants
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 91
participants
  Week 15, Adj M Phase, Improvement, n=91 | 51
  Week 15, Adj M Phase, No change, n=91 | 29
  Week 15, Adj M Phase, Deterioration, n=91 | 11
  Week 28, Adj O Phase, Improvement, n=21 | 17
  Week 28, Adj O Phase, No change, n=21 | 2
  Week 28, Adj O Phase, Deterioration, n=21 | 2
  Week 28, Mono Phase, Improvement, n=63 | 43
  Week 28, Mono Phase, No change, n=63 | 14
  Week 28, Mono Phase, Deterioration, n=63 | 6
  Week 28, WD, Improvement, n=35 | 7
  Week 28, WD, No change, n=35 | 12
  Week 28, WD, Deterioration, n=35 | 16

7. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure (BP) at the Indicated Time Points in the Study
Description: Change from Baseline was calculated by subtracting the values of systolic and diastolic blood pressures recorded by the investigator at the indicated time points in the study from the respective Baseline values.
Time Frame: Baseline (Week 0) and Week 15 (Adj M Phase), Week 28 (Adj O Phase), Week 28 (Mono Phase), Week 28 (WD), and Week 30/33 (End of study [EOS])
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 119
Millimeters of mercury
  Systolic BP, Week 15, Adj M Phase, n=88 | 1.51 (19.038)
  Systolic BP, Week 28, Adj O Phase, n=21 | -0.62 (15.377)
  Systolic BP, Week 28, Mono Phase, n=63 | 0.68 (20.509)
  Systolic BP, Week 28, WD, n=35 | -4.00 (15.566)
  Systolic BP, Week 30/33, EOS, n=119 | -2.19 (15.928)
  Diastolic BP, Week 15, Adj M Phase, n=88 | -1.22 (10.547)
  Diastolic BP, Week 28, Adj O Phase, n=21 | -1.05 (7.214)
  Diastolic BP, Week 28, Mono Phase, n=63 | -0.08 (10.754)
  Diastolic BP, Week 28, WD, n=35 | -2.09 (8.763)
  Diastolic BP, Week 30/33, EOS, n=119 | -2.07 (9.102)

8. Secondary Outcome: Change From Baseline in the Height at the Indicated Time Points in the Study
Description: Change from Baseline was calculated by subtracting the value of height measured by the investigator at the indicated time points in the study from the Baseline value.
Time Frame: as for outcome 7
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 120
centimeters
  Week 15, Adj M Phase, n=90 | 0.03 (1.302)
  Week 28, Adj O Phase, n=21 | 0.29 (2.217)
  Week 28, Mono Phase, n=62 | -0.03 (1.293)
  Week 28, WD, n=36 | -0.03 (1.028)
  Week 30/33, EOS, n=120 | 0.03 (1.417)

9. Secondary Outcome: Change From Baseline in the Weight at the Indicated Time Points in the Study
Description: Change from Baseline was calculated by subtracting the value of weight measured by the investigator at the indicated time points in the study from the Baseline value.
Time Frame: as for outcome 7
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 119
kilograms
  Week 15, Adj M Phase, n=88 | -0.22 (3.204)
  Week 28, Adj O Phase, n=21 | -0.41 (2.968)
  Week 28, Mono Phase, n=62 | -0.48 (3.520)
  Week 28, WD, n=36 | -0.27 (3.735)
  Week 30/33, EOS, n=119 | -0.41 (3.470)

10. Secondary Outcome: Change From Baseline in the Basophil, Eosinophil, Hemoglobin, Lymphocyte, Monocyte, Absolute Neutrophil Count (ANC), Platelet Count, and White Blood Cell (WBC) Count at the Indicated Time Points in the Study
Description: The blood samples collected at the study visits were analyzed and assessed at the central laboratory, and the investigator reviewed and assessed the clinical significance. Change from Baseline was calculated by subtracting the value of basophil, eosinophil, hemoglobin, lymphocyte, monocyte, ANC, platelet count, and WBC count at the indicated time points in the study from the Baseline value.
Time Frame: Baseline (Week 0) and Week 15 (Adj M Phase), Week 28 (Adj O Phase), Week 28 (Mono Phase), and Week 28 (WD)
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Median (Full Range); unit: Giga (10^9) cells per liter
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 89
Giga (10^9) cells per liter
  Basophil, Week 15, Adj M, n=85 | 0.00 [-0.03 to 0.06]
  Basophil, Week 28, Adj O, n=19 | 0.00 [-0.02 to 0.02]
  Basophil, Week 28, Mono, n=55 | 0.00 [-0.05 to 0.05]
  Basophil, Week 28, WD, n=33 | 0.00 [-0.04 to 0.04]
  Eosinophil, Week 15, Adj M, n=89 | 0.00 [-0.38 to 0.55]
  Eosinophil, Week 28, Adj O, n=21 | 0.01 [-0.06 to 0.26]
  Eosinophil, Week 28, Mono, n=61 | 0.01 [-0.23 to 0.54]
  Eosinophil, Week 28, WD, n=33 | -0.01 [-0.17 to 0.84]
  Hemoglobin, Week 15, Adj M, n=85 | -4.00 [-38.00 to 19.00]
  Hemoglobin, Week 28, Adj O, n=19 | -6.00 [-22.00 to 4.00]
  Hemoglobin, Week 28, Mono, n=55 | -4.00 [-25.00 to 10.00]
  Hemoglobin, Week 28, WD, n=33 | -2.00 [-21.00 to 31.00]
  Lymphocytes, Week 15, Adj M, n=85 | -0.12 [-1.55 to 1.52]
  Lymphocytes, Week 28, Adj O, n=19 | -0.05 [-0.61 to 0.40]
  Lymphocytes, Week 28, Mono, n=55 | -0.20 [-1.75 to 0.62]
  Lymphocytes, Week 28, WD, n=33 | -0.09 [-0.94 to 0.66]
  Monocytes, Week 15, Adj M, n=85 | -0.03 [-0.41 to 0.47]
  Monocytes, Week 28, Adj O, n=19 | 0.00 [-0.55 to 0.26]
  Monocytes, Week 28, Mono, n=55 | -0.04 [-0.37 to 0.40]
  Monocytes, Week 28, WD, n=33 | -0.01 [-0.48 to 0.64]
  Absolute Neutrophil Count, Week 15, Adj M, n=85 | -0.23 [-3.00 to 5.04]
  Absolute Neutrophil Count, Week 28, Adj O, n=19 | 0.09 [-2.17 to 3.31]
  Absolute Neutrophil Count, Week 28, Mono, n=55 | -0.17 [-3.18 to 2.71]
  Absolute Neutrophil Count, Week 28, WD, n=33 | 0.17 [-1.99 to 6.47]
  Platelet Count, Week 15, Adj M, n=84 | 1.50 [-91.00 to 226.00]
  Platelet Count, Week 28, Adj O, n=19 | 3.00 [-55.00 to 216.00]
  Platelet Count, Week 28, Mono, n=54 | 0.00 [-75.00 to 104.00]
  Platelet Count, Week 28, WD, n=32 | 6.50 [-80.00 to 172.00]
  White Blood Cell Count, Week 15, Adj M, n=85 | -0.30 [-2.80 to 5.70]
  White Blood Cell Count, Week 28, Adj O, n=19 | -0.20 [-2.40 to 3.20]
  White Blood Cell Count, Week 28, Mono, n=55 | -0.60 [-3.50 to 2.00]
  White Blood Cell Count, Week 28, WD, n=33 | 0.30 [-2.20 to 6.00]

11. Secondary Outcome: Percent Change From Baseline in the Basophil, Eosinophil, Hemoglobin, Lymphocyte, Monocyte, Absolute Neutrophil Count, Platelet Count, and White Blood Cell Count at the Indicated Time Points in the Study
Description: The blood samples collected at the study visits were analyzed and assessed at the central laboratory, and the investigator reviewed and assessed the clinical significance. Percent change from Baseline = (value at each indicated time point in the study minus respective Baseline value divided by Baseline value) x 100.
Time Frame: Baseline (Week 0) and Week 15 (Adj M Phase), Week 28 (Adj O Phase), Week 28 (Mono Phase), and Week 28 (WD)
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Median (Full Range); unit: Percent change in counts
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 89
Percent change in counts
  Basophil, Week 15, Adj M, n=89 | 0.00 [-0.80 to 1.00]
  Basophil, Week 28, Adj O, n=21 | 0.00 [-0.50 to 0.50]
  Basophil, Week 28, Mono, n=61 | 0.00 [-0.80 to 0.90]
  Basophil, Week 28, WD, n=33 | 0.00 [-0.50 to 0.90]
  Eosinophil, Week 15, Adj M, n=89 | 0.20 [-4.40 to 10.90]
  Eosinophil, Week 28, Adj O, n=21 | 0.10 [-1.50 to 4.30]
  Eosinophil, Week 28, Mono, n=61 | 0.30 [-3.30 to 10.80]
  Eosinophil, Week 28, WD, n=33 | -0.20 [-2.90 to 17.60]
  Hematocrit, Week 15, Adj M, n=85 | -0.01 [-0.11 to 0.06]
  Hematocrit, Week 28, Adj O, n=19 | -0.02 [-0.07 to 0.02]
  Hematocrit, Week 28, Mono, n=55 | -0.01 [-0.09 to 0.04]
  Hematocrit, Week 28, WD, n=33 | -0.00 [-0.04 to 0.10]
  Lymphocytes, Week 15, Adj M, n=89 | -2.10 [-25.80 to 18.90]
  Lymphocytes, Week 28, Adj O, n=21 | -2.40 [-16.00 to 13.60]
  Lymphocytes, Week 28, Mono, n=61 | -1.50 [-23.90 to 12.40]
  Lymphocytes, Week 28, WD, n=33 | -1.60 [-14.20 to 8.10]
  Monocytes, Week 15, Adj M, n=89 | 0.00 [-8.90 to 6.50]
  Monocytes, Week 28, Adj O, n=21 | 0.10 [-10.90 to 5.10]
  Monocytes, Week 28, Mono, n=61 | -0.20 [-6.40 to 9.50]
  Monocytes, Week 28, WD, n=33 | -0.30 [-8.00 to 8.10]
  Total Neutrophils, Week 15, Adj M, n=89 | 1.3 [-26.30 to 30.40]
  Total Neutrophils, Week 28, Adj O, n=21 | 0.50 [-13.80 to 16.80]
  Total Neutrophils, Week 28, Mono, n=61 | 0.50 [-13.80 to 24.20]
  Total Neutrophils, Week 28, WD, n=33 | 1.20 [-12.00 to 19.20]

12. Secondary Outcome: Change From Baseline in the Mean Corpuscle Hemoglobin Concentration (MCHC), Albumin, and Total Protein at the Indicated Time Points in the Study
Description: The blood samples collected at the study visits were analyzed and assessed at the central laboratory, and the investigator reviewed and assessed the clinical significance. Change from Baseline was calculated by subtracting the values of MCHC, albumin, and total protein at the indicated time points in the study from the respective Baseline values.
Time Frame: Baseline (Week 0) and Week 15 (Adj M Phase), Week 28 (Adj O Phase), Week 28 (Mono Phase), and Week 28 (WD)
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Median (Full Range); unit: grams per liter
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 87
grams per liter
  MCHC, Week 15, Adj M, n=85 | -4.00 [-30.00 to 27.00]
  MCHC, Week 28, Adj O, n=21 | 1.00 [-18.00 to 26.00]
  MCHC, Week 28, Mono, n=61 | -5.00 [-31.00 to 24.00]
  MCHC, Week 28, WD, n=33 | 1.00 [-25.00 to 15.00]
  Albumin, Week 15, Adj M, n=87 | 0.00 [-5.00 to 7.00]
  Albumin, Week 28, Adj O, n=20 | -1.00 [-8.00 to 3.00]
  Albumin, Week 28, Mono, n=61 | 0.00 [-6.00 to 6.00]
  Albumin, Week 28, WD, n=33 | 0.00 [-9.00 to 6.00]
  Total Protein, Week 15, WD, n=87 | -1.0 [-13.0 to 8.0]
  Total Protein, Week 28, WD, n=20 | -3.00 [-11.0 to 3.0]
  Total Protein, Week 28, WD, n=61 | -1.0 [-15.0 to 6.0]
  Total Protein, Week 28, WD, n=33 | -1.0 [-15.0 to 7.0]

13. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin (MCH) at the Indicated Time Points in the Study
Description: The blood samples collected at the study visits were analyzed and assessed at the central laboratory, and the investigator reviewed and assessed the clinical significance. Change from Baseline was calculated by subtracting the value of MCH at the indicated time points in the study from the Baseline value.
Time Frame: Baseline (Week 0) and Week 15 (Adj M Phase), Week 28 (Adj O Phase), Week 28 (Mono Phase), and Week 28 (WD)
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Median (Full Range); unit: picograms
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 85
picograms
  Week 15, Adj M, n=85 | -0.10 [-3.30 to 2.60]
  Week 28, Adj O, n=19 | 0.10 [-1.20 to 1.60]
  Week 28, Mono, n=55 | -0.20 [-2.30 to 1.40]
  Week 28, WD, n=33 | -0.20 [-1.90 to 3.50]

14. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume (MCV) at the Indicated Time Points in the the Study
Description: The blood samples collected at the study visits were analyzed and assessed at the central laboratory, and the investigator reviewed and assessed the clinical significance. Change from Baseline was calculated by subtracting the value of MCV at the indicated time points in the study from the Baseline value.
Time Frame: Baseline (Week 0) and Week 15 (Adj M Phase), Week 28 (Adj O Phase), Week 28 (Mono Phase), and Week 28 (WD)
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Median (Full Range); unit: Femtoliters
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 85
Femtoliters
  Week 15, Adj M, n=85 | 0.00 [-7.00 to 9.00]
  Week 28, Adj O, n=19 | -1.00 [-7.00 to 5.00]
  Week 28, Mono, n=55 | 1.00 [-9.00 to 7.00]
  Week 28, WD, n=33 | 0.00 [-4.00 to 12.00]

15. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) Count at the Indicated Time Points in the Study
Description: The blood samples collected at the study visits were analyzed and assessed at the central laboratory, and the investigator reviewed and assessed the clinical significance. Change from Baseline was calculated by subtracting the value of RBC count at the indicated time points in the study from the Baseline value. Change from baseline is measured as the number of red blood cells x 10^12 per liter.
Time Frame: Baseline (Week 0) and Week 15 (Adj M Phase), Week 28 (Adj O Phase), Week 28 (Mono Phase), and Week 28 (WD)
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Median (Full Range); unit: Tera (10^12) cells per liter
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 85
Tera (10^12) cells per liter
  Week 15, Adj M, n=85 | -0.10 [-0.90 to 0.40]
  Week 28, Adj O, n=19 | -0.20 [-0.80 to 0.10]
  Week 28, Mono, n=55 | -0.10 [-0.70 to 0.40]
  Week 28, WD, n=33 | 0.00 [-0.50 to 1.00]

16. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (Alk P), Alanine Amino Transferase (Ala AT), and Aspartate Amino Transferase (Asp AT) at the Indicated Time Points in the Study
Description: The blood samples collected at the study visits were analyzed and assessed at the central laboratory, and the investigator reviewed and assessed the clinical significance. Change from Baseline was calculated by subtracting the value of Alk P, Ala AT, and Asp AT at the indicated time points in the study from the Baseline value.
Time Frame: Baseline (Week 0) and Week 15 (Adj M Phase), Week 28 (Adj O Phase), Week 28 (Mono Phase), and Week 28 (WD)
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Median (Full Range); unit: International units per liter
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 89
International units per liter
  Alk P, Week 15, Adj M, n=87 | 1.00 [-86.0 to 141.00]
  Alk P, Week 28, Adj O, n=20 | -0.50 [-72.0 to 20.0]
  Alk P, Week 28, Mono, n=61 | -5.0 [-118.0 to 49.0]
  Alk P, Week 28, WD, n=33 | 2.00 [-90.0 to 90.00]
  Ala-AT Week 15, Adj M, n=87 | -2.00 [-30.0 to 71.0]
  Ala-AT, Week 28, Adj O, n=20 | -1.0 [-10.0 to 23.0]
  Ala-AT, Week 28, Mono, n=61 | -2.0 [-32.0 to 55.0]
  Ala-AT, Week 28, WD, n=33 | -2.0 [-20.0 to 7.0]
  Asp-AT, Week 15, Adj M, n=87 | -1.0 [-19.0 to 47.0]
  Asp-AT, Week 28, WD, n=32 | -3.0 [-34.0 to 7.0]
  Asp-AT, Week 28, Adj O, n=20 | -2.0 [-13.0 to 18.0]
  Asp-AT, Week 28, Mono, n=60 | 0.00 [-15.0 to 17.0]

17. Secondary Outcome: Change From Baseline in Direct Bilirubin (DB), Total Bilirubin (TB), and Creatinine at the Indicated Time Points in the Study
Description: The blood samples collected at the study visits were analyzed and assessed at the central laboratory, and the investigator reviewed and assessed the clinical significance. Change from Baseline was calculated by subtracting the value of DB, TB, and creatinine at the indicated time points in the study from the Baseline value.
Time Frame: Baseline (Week 0) and Week 15 (Adj M Phase), Week 28 (Adj O Phase), Week 28 (Mono Phase), and Week 28 (WD)
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Median (Full Range); unit: micromoles (µmol) per liter
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 88
micromoles (µmol) per liter
  DB, Week 15, Adj M, n=87 | 0.0 [-1.7 to 6.8]
  DB, Week 28, Adj O, n=20 | 0.0 [-3.4 to 1.7]
  DB, Week 28, Mono, n=61 | 0.0 [-1.7 to 12.0]
  DB, Week 28, WD, n=33 | 0.0 [-1.7 to 1.7]
  TB, Week 15, Adj M, n=88 | 0.0 [-8.6 to 15.4]
  TB, Week 28, Adj O, n=20 | 0.0 [-3.4 to 1.7]
  TB, Week 28, Mono, n=61 | 1.7 [-8.6 to 12.0]
  TB, Week 28, WD, n=33 | 0.0 [-3.4 to 5.1]
  Creatinine, Week 15, Adj M, n=88 | 8.8 [-17.7 to 53.0]
  Creatinine, Week 28, Adj O, n=20 | 8.8 [0.0 to 203.3]
  Creatinine, Week 28, Mono, n=61 | 8.8 [-17.7 to 53.0]
  Creatinine, Week 28, WD, n=33 | 0.0 [-17.7 to 17.7]

18. Secondary Outcome: Change From Baseline in Cholesterol, High Density Lipoprotein (HDL) Cholesterol, Low Density Lipoprotein (LDL) Cholesterol, Glucose, Potassium, Sodium, Triglycerides, and Urea/Blood Urea Nitrogen (BUN) at the Indicated Time Points
Description: The blood samples collected at the study visits were analyzed and assessed at the central laboratory, and the investigator reviewed and assessed the clinical significance. Change from Baseline was calculated by subtracting the value of cholesterol, HDL cholesterol, LDL cholesterol, glucose, potassium, sodium, triglycerides, and urea/BUN at the indicated time points in the study from the Baseline value.
Time Frame: Baseline (Week 0) and Week 15 (Adj M Phase), Week 28 (Adj O Phase), Week 28 (Mono Phase), and Week 28 (WD)
Population: Safety Population. Only those participants with both a baseline and post-baseline value were analyzed.
Measure: Median (Full Range); unit: millimoles (mmol) per liter
Arm/Group | LTG-XR Tablets
Number analyzed (Participants) | 87
millimoles (mmol) per liter
  Cholesterol, Week 15, Adj M, n=87 | -0.1 [-1.7 to 1.7]
  Cholesterol, Week 28, Adj O, n=20 | -0.1 [-2.2 to 0.9]
  Cholesterol, Week 28, Mono, n=61 | -0.3 [-2.5 to 1.2]
  Cholesterol, Week 28, WD, n=33 | -0.1 [-3.5 to 1.0]
  HDL Cholesterol, Week 15, Adj M, n=87 | 0.1 [-1.0 to 0.6]
  HDL Cholesterol, Week 28, Adj O, n=20 | -0.0 [-0.4 to 0.6]
  HDL Cholesterol, Week 28, Mono, n=61 | 0.0 [-0.7 to 0.7]
  HDL Cholesterol, Week 28, WD, n=33 | 0.1 [-0.9 to 0.4]
  LDL Cholesterol, Week 15, Adj M, n=86 | -0.0 [-1.1 to 1.2]
  LDL Cholesterol, Week 28, Adj O, n=19 | -0.2 [-1.9 to 1.1]
  LDL Cholesterol, Week 28, Mono, n=61 | -0.1 [-1.8 to 1.6]
  LDL Cholesterol, Week 28, WD, n=32 | -0.1 [-0.8 to 1.7]
  Glucose, Week 15, Adj M, n=87 | -0.1 [-5.8 to 5.3]
  Glucose, Week 28, Adj O, n=20 | 0.1 [-6.7 to 6.7]
  Glucose, Week 28, Mono, n=61 | 0.1 [-3.6 to 6.4]
  Glucose, Week 28, WD, n=33 | 0.3 [-5.2 to 4.2]
  Potassium, Week 15, Adj M, n=87 | 0.0 [-1.2 to 1.1]
  Potassium, Week 28, Adj O, n=20 | -0.1 [-0.7 to 1.2]
  Potassium, Week 28, Mono, n=60 | 0.0 [-1.3 to 1.2]
  Potassium, Week 28, WD, n=32 | 0.0 [-1.0 to 0.9]
  Sodium, Week 15, Adj M, n=87 | 0.0 [-4.0 to 6.0]
  Sodium, Week 28, Adj O, n=20 | 0.5 [-7.0 to 4.0]
  Sodium, Week 28, Mono, n=61 | -1.0 [-5.0 to 9.0]
  Sodium, Week 28, WD, n=33 | 1.0 [-3.0 to 7.0]
  Triglyceride, Week 28, WD, n=87 | -0.3 [-2.3 to 0.9]
  Triglyceride, Week 28, WD, n=20 | -0.1 [-1.7 to 1.6]
  Triglyceride, Week 28, WD, n=61 | -0.4 [-1.9 to 1.1]
  Triglyceride, Week 28, WD, n=33 | 1.0 [-4.6 to 1.1]
  Urea/BUN, Week 28, WD, n=87 | 0.0 [-10.4 to 5.4]
  Urea/BUN, Week 28, WD, n=20 | 0.5 [-2.1 to 13.2]
  Urea/BUN, Week 28, WD, n=61 | 0.0 [-6.4 to 6.8]
  Urea/BUN, Week 28, WD, n=33 | 0.4 [-4.3 to 3.6]

19. Secondary Outcome: Serum LTG Concentrations at Different LTG Doses Based on the Concomitant AED Groups: Neutral (Without Known Enzyme-inducing AED [EIAED], Valproate [VPA]) With EIAED, and With VPA
Description: The blood samples were collected at the specified study visits; however, serum LTG concentrations were summarized by dose regimen, not by study week. The serum was assayed for LTG using an approved method under the management of Worldwide Bioanalysis, GlaxoSmithKline.
Time Frame: Weeks 4, 7, 11, 15, 20, 24, and 28
Population: Safety Population. Participants with missing data were not analyzed. Not all participants received all doses at each blood draw; therefore, participants were only analyzed for the dose received at blood draw.
Measure: Median (Full Range); unit: Micrograms per milliliter
Units Other Than Participants: serum concentrations
Groups:
- LTG-XR + Neutral: LTG-XR tablets (25, 50, 100, and 200 mg) were administered OD in the 7-week (w) Dose-Escalation Phase and titrated to target doses of 300, 500, or 200 mg/day for participants (par.) depending on their concomitant AED (does not include VPA or EIAEDs), followed by an 8-w Adjunctive Maintenance Phase in which LTG-XR tablets were administered OD at the target dose. Par. on a single concomitant AED who converted to LTG-XR monotherapy (based on investigator's judgment) entered the 5-w Conversion Phase, followed by an 8-w Monotherapy Phase, whereas par. who did not transition to monotherapy entered the 13-w Adjunctive Optimization Phase. At the end of the study, par. entered the 2- to 5-w Taper/Follow-Up Phase, in which par. either switched to commercial LTG (received same total daily dose of commercial LTG in 2 divided doses [BID]) or did not switch to commercial LTG (current dose was reduced by approximately one-fourth per week) with a final visit 2 weeks after last LTG-XR dose.
- LTG-XR + EIAEDs: LTG-XR tablets (25, 50, 100, and 200 mg) were administered OD in the 7-w Dose-Escalation Phase and titrated to target doses of 300, 500, or 200 mg/day for participants (par.) depending on their concomitant AED (included EIAEDs), followed by an 8-w Adjunctive Maintenance Phase in which LTG-XR tablets were administered OD at the target dose. Par. on a single concomitant AED who converted to LTG-XR monotherapy (based on investigator's judgment) entered the 5-w Conversion Phase, followed by an 8-w Monotherapy Phase, whereas par. who did not transition to monotherapy entered the 13-w Adjunctive Optimization Phase. At the end of the study, par. entered the 2- to 5-w Taper/Follow-Up Phase, in which par. either switched to commercial LTG (received same total daily dose of commercial LTG in 2 divided doses [BID]) or did not switch to commercial LTG (current dose was reduced by approximately one-fourth per week) with a final visit 2 weeks after last LTG-XR dose.
- LTG-XR + VPA: LTG-XR tablets (25, 50, 100, and 200 mg) were administered OD in the 7-w Dose-Escalation Phase and titrated to target doses of 300, 500, or 200 mg/day for participants (par.) depending on their concomitant AED (included VPA), followed by an 8-w Adjunctive Maintenance Phase: LTG-XR tablets administered OD at the target dose. Par. on a single concomitant AED who converted to LTG-XR monotherapy (based on investigator's judgment) entered the 5-w Conversion Phase, followed by an 8-w Monotherapy Phase, whereas par. who did not transition to monotherapy entered the 13-w Adjunctive Optimization Phase. At the end of the study, par. entered the 2- to 5-w Taper/Follow-Up Phase, in which par. either switched to commercial LTG (received same total daily dose of commercial LTG in 2 divided doses [BID]) or did not switch to commercial LTG (current dose was reduced by approximately one-fourth per week) with a final visit 2 weeks after last LTG-XR dose.
Arm/Group | LTG-XR + Neutral | LTG-XR + EIAEDs | LTG-XR + VPA
Number analyzed (Participants) | 87 | 50 | 12
Number analyzed (serum concentrations) | 439 | 243 | 54
Micrograms per milliliter
  12.5 mg, n=0, 0, 1 | NA [NA to NA] — No dose was given for this regimen. | NA [NA to NA] — No dose was given for this regimen. | 0.957 [NA to NA] — No full range is provided for the median value because only one participant was analyzed.
  25 mg, n=0, 0, 8 | NA [NA to NA] — No dose was given for this regimen. | NA [NA to NA] — No dose was given for this regimen. | 1.362 [0.817 to 2.885]
  50 mg, n=30, 2, 8 | 1.281 [0.437 to 3.491] | 0.731 [0.727 to 0.734] | 2.972 [0.937 to 3.553]
  100 mg, n=40, 32, 6 | 3.425 [0.717 to 5.825] | 1.165 [0.442 to 4.254] | 4.723 [3.870 to 6.419]
  150 mg, n=11, 0, 6 | 5.653 [2.514 to 9.693] | NA [NA to NA] — No participants were analyzed in this group at this dose level. | 6.829 [3.549 to 10.804]
  200 mg, n=74, 22, 25 | 5.499 [1.449 to 12.926] | 1.583 [0.455 to 3.542] | 5.350 [3.301 to 13.750]
  225 mg, n=3, 0, 0 | 5.631 [4.815 to 5.642] | NA [NA to NA] — No participants were analyzed in this group at this dose level. | NA [NA to NA] — No participants were analyzed in this group at this dose level.
  250 mg, n=18, 11, 0 | 5.059 [2.329 to 10.969] | 4.073 [2.184 to 8.768] | NA [NA to NA] — No participants were analyzed in this group at this dose level.
  300 mg, n=193, 5, 0 | 5.493 [1.620 to 13.335] | 2.837 [1.898 to 3.558] | NA [NA to NA] — No participants were analyzed in this group at this dose level.
  350 mg, n=0, 3, 0 | NA [NA to NA] — No dose was given for this regimen. | 4.084 [3.794 to 4.165] | NA [NA to NA] — No participants were analyzed in this group at this dose level.
  400 mg, n=19, 46, 0 | 7.322 [2.899 to 13.843] | 4.012 [1.459 to 9.675] | NA [NA to NA] — No participants were analyzed in this group at this dose level.
  450 mg, n=0, 1, 0 | NA [NA to NA] — No dose was given for this regimen. | 2.975 [NA to NA] — No full range is provided for the median value because only one participant was analyzed. | NA [NA to NA] — No participants were analyzed in this group at this dose level.
  500 mg, n=51, 121, 0 | 6.994 [0.931 to 13.412] | 3.974 [0.905 to 11.451] | NA [NA to NA] — No participants were analyzed in this group at this dose level.

20. Secondary Outcome: Apparent Clearance (CL/F) Based on the Concomitant AED Groups: Neutral, With EIAED, and With VPA
Description: Individual serum LTG concentration data were subjected to population pharmacokinetic methodologies based on the concomitant AED groups. Clearance is defined as the volume of LTG per unit time eliminated from serum. Serum LTG concentration-time data files incorporating, where appropriate, records of LTG administration, participant demography, and concomitant medication were supplied to Clinical Pharmacokinetics Modelling and Simulation, Clinical Pharmacology, and Discovery Medicine (CPDM) by Clinical Data Management as NONMEM compatible .csv files.
Time Frame: Weeks 4, 7, 11, 15, 20, 24, and 28
Population: as for outcome 19
Measure: Mean (95% Confidence Interval); unit: Liters per hour
Arm/Group | LTG-XR + Neutral | LTG-XR + EIAEDs | LTG-XR + VPA
Number analyzed (Participants) | 87 | 50 | 12
Liters per hour | 1.91 [1.73 to 2.09] | 2.07 [1.69 to 2.46] | -0.698 [-0.96 to -0.441]

21. Secondary Outcome: Apparent Volume of Distribution (V/F) for Participants in All Concomitant AED Groups Combined: Neutral, With EIAED, and With VPA
Description: Individual serum LTG concentration data were subjected to population pharmacokinetic methodologies based on the concomitant AED groups. V/F is defined as the apparent volume in which a drug is distributed immediately after it has been injected intravenously and equilibrated between plasma and the surrounding tissues. Serum LTG concentration-time data files incorporating, where appropriate, records of LTG administration, participant demography, and concomitant medication were supplied to CPDM by Clinical Data Management as NONMEM compatible .csv files.
Time Frame: Weeks 4, 7, 11, 15, 20, 24, and 28
Population: as for outcome 19
Measure: Mean (95% Confidence Interval); unit: liters
Groups:
- LTG-XR + Neutral, EIAEDs, and VPA: LTG-XR tablets (25, 50, 100, and 200 mg) were administered OD in the 7-week (w) Dose-Escalation Phase and titrated to target doses of 300, 500, or 200 mg/day for participants (par.) depending on their concomitant AED (included VPA and EIAEDs), followed by an 8-w Adjunctive Maintenance Phase in which LTG-XR tablets were administered OD at the target dose. Par. on a single concomitant AED who converted to LTG-XR monotherapy (based on investigator's judgment) entered the 5-w Conversion Phase, followed by an 8-w Monotherapy Phase, whereas par. who did not transition to monotherapy entered the 13-w Adjunctive Optimization Phase. At the end of the study, par. entered the 2- to 5-w Taper/Follow-Up Phase, in which par. either switched to commercial LTG (received same total daily dose of commercial LTG in 2 divided doses [BID]) or did not switch to commercial LTG (current dose was reduced by approximately one-fourth per week) with a final visit 2 weeks after last LTG-XR dose.
Arm/Group | LTG-XR + Neutral, EIAEDs, and VPA
Number analyzed (Participants) | 149
liters | 26.8 [7.40 to 46.6]

22. Secondary Outcome: Absorption Rate (KA) for Participants in All Concomitant AED Groups Combined: Neutral, With EIAED, and With VPA
Description: Individual serum LTG concentration data were subjected to population pharmacokinetic methodologies based on the concomitant AED groups. KA is defined as the rate at which a drug enters the body after administration. Serum LTG concentration-time data files incorporating, where appropriate, records of LTG administration, participant demography, and concomitant medication were supplied to CPDM by Clinical Data Management as NONMEM compatible .csv files.
Time Frame: Weeks 4, 7, 11, 15, 20, 24, and 28
Population: as for outcome 19
Measure: Mean (95% Confidence Interval); unit: 1/h
Arm/Group | LTG-XR + Neutral, EIAEDs, and VPA
Number analyzed (Participants) | 149
1/h | 0.0325 [0.0105 to 0.0549]

ADVERSE EVENTS:
Arm/Group | LTG-XR Tablets
Serious Adverse Events (participants affected / at risk) | 22/121
Other Adverse Events (participants affected / at risk) | 98/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LTG-XR Tablets (N=121)
Hip fracture (Injury, poisoning and procedural complications) | 3
Ataxia (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 2
Status epilepticus (Nervous system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Balance disorder (Nervous system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diverticulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Grand mal convulsion (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Lethargy (Nervous system disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 1
Thrombosis (Vascular disorders) | 1
Toxic encephalopathy (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LTG-XR Tablets (N=121)
Dizziness (Nervous system disorders) | 31
Balance disorder (Nervous system disorders) | 25
Fall (Injury, poisoning and procedural complications) | 22
Headache (Nervous system disorders) | 21
Tremor (Nervous system disorders) | 20
Fatigue (Nervous system disorders) | 17
Nausea (Gastrointestinal disorders) | 17
All rash (Skin and subcutaneous tissue disorders) | 14
Ataxia (Nervous system disorders) | 14
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 11
Pain In extremity (Musculoskeletal and connective tissue disorders) | 11
Gait disturbance (Nervous system disorders) | 10
Somnolence (Nervous system disorders) | 10
Arthralgia (Nervous system disorders) | 9
Confusional state (Nervous system disorders) | 8
Constipation (Gastrointestinal disorders) | 8
Decreased appetite (Gastrointestinal disorders) | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 7
Skin laceration (Skin and subcutaneous tissue disorders) | 7
Urinary tract infection (Renal and urinary disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.